CLINICAL TRIAL: NCT06443489
Title: A Phase I ,Open-label, Multicenter Clinical Study to Evaluate the Safety, Tolerability , Pharmacokinetics and Efficacy of SHR-4849 in Patients With Advanced Solid Tumors
Brief Title: A Trial of SHR-4849 in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-4849-101
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2024-05

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-4849 (Experimental)
  Interventions: Drug: SHR-4849

INTERVENTIONS:
Drug: SHR-4849 — SHR-4849

SUMMARY:
The study is being conducted to evaluate the safety, tolerability and efficacy of SHR-4849 injection in Advanced Solid Tumors. To explore the reasonable dosage of SHR-4849 for Advanced Solid Tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided informed consent prior to initiation of any study-procedures
2. Age from 18 to 75 years old at the time of signing the informed consent
3. Histologically or cytologically confirmed advanced solid tumors
4. At least one measurable lesion was identified per RECIST 1.1
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
6. Has a life expectancy of at least 3 months.
7. Adequate organ function
8. Subjects of both genders of child-bearing potential were required to use highly effective contraception from the time they provided written informed consent until 6 months after the last dose of the trial drug

Exclusion Criteria:

1. Subjects with active central nervous system (CNS) metastasis.
2. Subjects with a history of malignant tumors within 5 years prior to the first dose
3. Subjects with uncontrolled cancer pain.
4. Subjects with severe cardiovascular disease.
5. Subjects with clinically significant hemorrhage
6. Subjects with uncontrolled pleural effusion, peritoneal effusion and pericardial effusion
7. Subjects highly suspected of interstitial lung disease
8. Subjects with serious infection within 4 weeks prior to the first dose
9. Known history of human immunodeficiency virus (HIV)，active hepatitis B virus or hepatitis C virus infection.
10. The adverse events of previous antineoplastic therapy did not recover to NCI-CTCAE≤ grade 1
11. Subjects who received anti-cancer treatment within 4 weeks prior to the first dose
12. Subjects who received major surgery within 4 weeks prior to the first dose
13. Subjects who plan to receive or have received live vaccines within 28 days prior to the first dose.
14. Female subjects who were pregnant, lactating, or planned to become pregnant during the study period
15. Known allergic to any component of SHR-4849 products
16. Alcohol abuse, drug abuse, other serious medical conditions (including mental illness) requiring combined treatment, and other conditions that may affect subject safety or data collection.
17. Based on the investigator's judgment, subjects with other conditions that may affect study results, interfere with study procedures,

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
DLT：the incidence of events associated with the investigational drug determined by the investigator during the observation period | up to 21 days
Incidence and severity of AE/SAE：According to NCI-CTCAE v5.0 evaluation criteria, from the signing of informed consent to the end of safety follow-up； | up to 24 months
MTD or MAD：after all subjects of dose escalation phase be enrolled，and all subjects complete at least one cycle of dosing observation. | up to 24 months
RP2D：after all subjects of dose escalation and dose expansion phase be enrolled，and all subjects complete at least one cycle of dosing observation. | up to 24 months

SECONDARY OUTCOMES:
ORR： Objective Response Rate (ORR) as Assessed by investigators. The proportion of subjects whose best response was PR or CR according to RECIST1.1 | up to 24 months
DCR：Disease Control Rate(DCR) as Assessed by investigators. the proportion of subjects whose best response was PR or CR or SD according to RECIST1.1 | up to 24 months
DoR: Duration of Response (DOR) as Assessed by investigators according to RECIST1.1, Defined as the period of time from the first documented tumor response to the first documented objective progression or death of any cause. | up to 24 months
PFS: Progression-free Survival (PFS) as Assessed by investigators according to RECIST1.1. Defined as the time from the initiation of the first medication to tumor progression or death from any cause (whichever comes first)； | up to 24 months
OS: Overall Survival . Defined as the time from the initiation of the first medication to death from any cause. | up to 30 months

CONTACTS AND LOCATIONS:
Locations (1):
- Jilin Cancer Hospital, Jilin, Changchun, China

IPD SHARING:
Plan to Share IPD: Undecided